CLINICAL TRIAL: NCT00730795
Title: A Phase I Open Label, Dose-Escalation Study to Evaluate the Safety and Immunogenicity of the Recombinant Mycobacterium Tuberculosis Vaccine, Mtb72F With AS02A Adjuvant, When Administered Intramuscularly to Healthy PPD-Negative Adults
Brief Title: Safety and Immunogenicity of a Candidate Tuberculosis (TB) Vaccine Given to PPD-Negative Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Corixa Corporation (Industry)
Responsible Party: Isabelle Harpigny, GSK Biologicals
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 692342/001; CCTB001-01
Record Dates: First submitted 2008-08-07; First posted 2008-08-08 (Estimated); Last update posted 2008-08-08 (Estimated); Status verified 2008-08

CONDITIONS: Tuberculosis (TB)
Keywords: Tuberculosis vaccine
MeSH Terms: conditions — Tuberculosis

ARMS (2):
- Group A (Experimental): Subjects receiving the low-dose antigen candidate TB vaccine
  Interventions: Biological: GSK's candidate Mycobacterium tuberculosis vaccine 692342
- Group B (Experimental): Subjects receiving the high-dose antigen candidate TB vaccine
  Interventions: Biological: GSK's candidate Mycobacterium tuberculosis vaccine 692342

INTERVENTIONS:
Biological: GSK's candidate Mycobacterium tuberculosis vaccine 692342 — Intramuscular injection, 3 doses at 0, 1, 2 months Different antigen doses (low and high)

SUMMARY:
This Phase I study will evaluate the safety and immunogenicity of two doses GSK Biologicals' candidate TB vaccine (692342) according to a 0, 1, 2 months schedule in PPD-negative adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female between 18 and 40 years of age at the time of screening
* Negative PPD skin test at screening.
* Subjects must have chest X-ray showing no evidence of pulmonary pathology.
* Female subjects of childbearing potential must have a negative serum pregnancy test at screening, must not be breast-feeding and are required to use adequate contraception from enrolment till 1 month after dose 3.
* Screening laboratory values must be within the laboratory normal ranges.
* Negative for human immunodeficiency virus-1 and 2 (HIV 1/2) antibody, hepatitis B surface antigen (HBsAg), and hepatitis C virus (HCV) antibody.
* Subjects must give written informed consent.
* Subjects must be willing to make all evaluation visits, be readily reachable by telephone or personal contact by the study site personnel and have a permanent address.
* Subjects' resting seated vital signs must be within the protocol-defined ranges.

Exclusion Criteria:

* History of prior Bacillus Calmette-Guérin (BCG) vaccinations.
* History of documented exposure to Mycobacterium tuberculosis.
* History of previous administration of experimental Mycobacterium tuberculosis vaccines or previous exposure to experimental products containing components of the experimental vaccine.
* History of employment in a healthcare facility in a capacity that had direct or indirect contact with TB patients.
* Administration of any immunoglobulins or any immunotherapy within the 3 months preceding the first dose of study vaccination, and/or any blood products within the 4 months preceding HIV screening, or planned administrations during the study period.
* Use of St. John's Wort within six months of the Day 0 visit or planned administrations during the study period.
* Participation in another experimental protocol and/or receipt of any investigational products within 30 days prior to Day 0.
* History of autoimmune disease or causes of immunosuppressive states.
* History of any acute or chronic illness or medication that, in the opinion of the Investigator, may interfere with the evaluation of the safety or immunogenicity of the vaccine.
* History of significant psychiatric illness.
* Current drug or alcohol abuse
* History of previous anaphylaxis or severe allergic reaction to vaccines or any other allergen.
* Subjects who are, in the opinion of the investigator, at significantly increased risk of non-cooperation with requirements of the study protocol.
* Any chronic drug therapy to be continued during the study period, with the exception of vitamins and/or dietary supplements (including mineral preparations such as calcium carbonate), herbal medications except St. John's Wort, birth control pills, anti-histamines for seasonal allergies, SSRIs (e.g. Prozac, Zoloft, Paxil), NSAIDs (e.g. aspirin, ibuprofen), and acetominophen.
* Chronic administration (defined as more than 14 days total) of immunosuppressants or other immune modifying drugs within six months prior to the first vaccine dose.
* History of chronic or intermittently recurring illnesses such as migraine headaches, diabetes, heart disease, and asthma.
* Current administration of anti-TB prophylaxis or therapy.
* History of administration of a live attenuated virus vaccine within 30 days of enrollment.
* History of administration of a subunit or killed vaccine within 14 days of enrollment.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2004-01; Primary Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Occurrence of dose limiting toxicity | From study start up to Day 56.
Occurrence of serious adverse events | During the entire study period.
Occurrence of adverse events | At each visit
Laboratory measurements of serum chemistry and hematology | At study start, prior to each vaccination and 1 and 6 months after dose 3
Resting vital signs (blood pressure, pulse, temperature) | At study start, prior to each vaccination and 1 and 6 months after dose 3
Chest X-ray findings | At study start and study end

SECONDARY OUTCOMES:
Evaluation of T cell and antibody responses to the fusion protein and to each of the three Mycobacterium tuberculosis antigen domains. | Prior to each vaccination and 1 and 6 months after dose 3
Evaluation of PPD skin reactivity | At study start and study end

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Clinical Trials Call Center, Tacoma, Washington, United States

REFERENCES:
- [Derived] Von Eschen K, Morrison R, Braun M, Ofori-Anyinam O, De Kock E, Pavithran P, Koutsoukos M, Moris P, Cain D, Dubois MC, Cohen J, Ballou WR. The candidate tuberculosis vaccine Mtb72F/AS02A: Tolerability and immunogenicity in humans. Hum Vaccin. 2009 Jul;5(7):475-82. doi: 10.4161/hv.8570. Epub 2009 Jul 27. PMID 19587528